CLINICAL TRIAL: NCT05058586
Title: The Effects of Aerobic Exercise Training on Cardiorespiratory Fitness, Functional Capacity, Balance and Ventricular Repolarization Indices in Stroke Patients
Brief Title: The Effects of Aerobic Exercise Training on Cardiorespiratory Fitness in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21
Record Dates: First submitted 2021-08-25; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Stroke, Cardiovascular
Keywords: underwater walking theraphy; anti-gravity treadmill training
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional theraphy group (Active Comparator): 13 patients received twenty sessions of conventional therapy for four weeks
  Interventions: Other: The Effects of Aerobic Exercise Training on Cardiorespiratory Fitness, Functional Capacity, Balance and Ventricular Repolarization Indices in Stroke Patients
- Anti gravity treadmill training (Active Comparator): 13 patients received twenty sessions of conventional therapy for four weeks and Alter-G training was performed 3 days/week for 4 weeks, with up to 30 min. of training per session.
  Interventions: Other: The Effects of Aerobic Exercise Training on Cardiorespiratory Fitness, Functional Capacity, Balance and Ventricular Repolarization Indices in Stroke Patients
- Underwater walking therapy group (Active Comparator): 13 patients received twenty sessions of conventional therapy for four weeks and three sessions of aerobic exercise treatment of 45 minutes per week underwater
  Interventions: Other: The Effects of Aerobic Exercise Training on Cardiorespiratory Fitness, Functional Capacity, Balance and Ventricular Repolarization Indices in Stroke Patients

INTERVENTIONS:
Other: The Effects of Aerobic Exercise Training on Cardiorespiratory Fitness, Functional Capacity, Balance and Ventricular Repolarization Indices in Stroke Patients — Seventy patients with history of stroke admitted to our center between July 2017 and January 2018. Subjects participated in the study were randomly assigned to anti-gravity treadmill training, underwater walking therapy and control group. We examined aerobic capacity of participants by using 6-minute walk test and cycle ergometer testing before starting the treatment along with one month follow up. Patient's balance examined by using the Berg Balance Scale (BBS).

SUMMARY:
Background:

Aerobic exercise training has favorable effects on quality of life, motor recovery, and aerobic endurance after stroke.

Objectives: In this study, the investigators aimed to explore the effects of anti-gravity treadmill gait training and underwater walking therapy on cardiorespiratory fitness in stroke survivors.

DETAILED DESCRIPTION:
Methods: Seventy patients with a history of stroke were admitted to our center between July 2017 and January 2018. Subjects who participated in the study were randomly assigned to anti-gravity treadmill training, underwater walking therapy, and control group. Investigators examined the aerobic capacity of participants by using the 6-minute walk test and cycle ergometer testing before starting the treatment along with a one-month follow-up. The patient's balance was examined by using the Berg Balance Scale (BBS).

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 80 and diagnosed with stroke and time from stroke onset to admission were longer than three months
* Independent walking ability more than 10 meters with or without assistance
* Patients whose cognitive and functional status were suitable for the training program

Exclusion Criteria:

* Had a previous history of stroke
* Bilateral hemiplegia
* Leg-length difference >2.0 cm
* Fixed flexion contracture or severe joint deformity
* Bladder or bowel incontinence
* Open wound
* Cardiovascular complaints and can not tolerate exercise training
* Other neurological comorbidities including, multiple sclerosis (MS), spinal cord injury (SCI), traumatic brain injury (TBI), Parkinson's disease, and intracranial tumors
* Congestive heart failure
* Atrial fibrillation (AF), use of antiarrhythmic drugs affecting QT duration, any type of bundle branch block on electrocardiogram (ECG)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | Change from baseline resting heart rate at 4 weeks
  Resting heart rate
6-minute walk test | Change from baseline maximum heart rate at 4 weeks
  Maximum heart rate
6-minute walk test | Change from baseline length of walking distance at 4 weeks
  Length of walking distance
Cycle ergometer training | Change from baseline maximum heart rate at 4 weeks
  Maximum heart rate
Cycle ergometer training | Change from baseline period of completion of test at 4 weeks
  Period of completion of test
Cycle ergometer training | Change from baseline METs scores at 4 weeks
  METs scores
Cycle ergometer training | Change from baseline VO2 max at 4 weeks
  VO2 max

OTHER OUTCOMES:
Echocardiographic parameters | Change from baseline LV ejection fraction at 4 weeks
  LV ejection fraction
Electrocardiographic parameters | Change from baseline QTc at 4 weeks
  QTc
Electrocardiographic parameters | Change from baseline Tp-e interval at 4 weeks
  Tp-e interval
Electrocardiographic parameters | Change from baseline Tp-e/ QT at 4 weeks
  Tp-e/ QT
Electrocardiographic parameters | Change from baseline Tp-e/QTc at 4 weeks
  Tp-e/QTc

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Konya City Hospital, Meram, Konya
  - Gaziler Physical Theraphy and Rehabilitation, Ankara

IPD SHARING:
Plan to Share IPD: No